CLINICAL TRIAL: NCT02533466
Title: Study to Investigate the Initial Stages of Enamel Erosion in Vivo
Brief Title: In Vivo Investigation of Initial Stages of Enamel Erosion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 204739
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-03

CONDITIONS: Tooth Erosion
MeSH Terms: conditions — Tooth Erosion | interventions — Sodium Fluoride; potassium nitrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): Subjects will apply a full ribbon of dentifrice and brush their teeth for 1 timed minute using a wetted toothbrush, swish the resulting slurry around the mouth for 30 seconds making sure it contacts the selected teeth, spit out slurry and rinse mouth for 10 seconds with water.
  Interventions: Other: Sodium fluoride + potassium nitrate
- Reference Product (Placebo Comparator): Subjects will apply a full ribbon of dentifrice and brush their teeth for 1 timed minute using a wetted toothbrush, swish the resulting slurry around the mouth for 30 seconds making sure it contacts the selected teeth, spit out slurry and rinse mouth for 10 seconds with water.
  Interventions: Other: Potassium nitrate

INTERVENTIONS:
Other: Sodium fluoride + potassium nitrate — Marketed toothpaste containing 1450ppm fluoride as sodium fluoride and 5% potassium nitrate
  Arms: Test Product
Other: Potassium nitrate — Experimental toothpaste containing 5% potassium nitrate
  Arms: Reference Product

SUMMARY:
This exploratory study is designed to help develop a clinical model to measure the earlier stages of dietary acid medicated enamel loss. The study will use fluoride as positive control to explore the validity of this design.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged at least 18 years
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon oral examination.
* Absence of any condition that would impact the participant's safety or well-being, or affect the participant's ability to understand and follow study procedures and requirements.
* Two anterior maxillary teeth, without signs of toothwear or exposed dentine, facial restorations, abutments for fixed or removable partial dentures, full crowns or veneers, orthodontic bands or cracked enamel that would interfere with the study evaluations.

Exclusion Criteria:

* Pregnant or breast feeding women
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Recent history (within the last year) of alcohol or other substance abuse
* Presence of a disease or medication which in the opinion of the investigator, will impact on assessments
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening
* Surface irregularities, discoloration due to trauma, restorations and hypo or hyperplasic areas which, in the opinion of the investigator or dental assessor, would prevent accurate impressions and grading
* Daily doses of a medication which, in the opinion of the investigator, could impact the assessment, for example acidic medications
* Any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10-01; Primary Completion 2015-11-06 (Actual); Study Completion 2015-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bristol, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 1 center in United Kingdom.
Pre-assignment Details: A total of 30 participants were screened and all of them were randomized.
Groups:
- Test Product; Reference Product: Participants applied a full ribbon of dentifrice and brushed their teeth for 1 timed minute using a wet toothbrush, swished the resulting slurry around the mouth for 30 seconds making sure it contacted the selected teeth, spitted out slurry and rinsed mouth for 10 seconds with water.
Period: Overall Study
Arm/Group | Test Product | Reference Product
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Per Protocol (PP) population was the primary population.
Groups:
- Test Product: Participants applied a full ribbon of dentifrice and brushed their teeth for 1 timed minute using a wet toothbrush and swished the resulting slurry around the mouth for 30 seconds making sure it contacted the selected teeth, spitted out slurry and rinsed mouth for 10 seconds with water.
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (11.17) | 38.1 (12.21) | 37.1 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-acid Challenge (Baseline) Tooth Impression Grading Score Immediately Following an Acid Challenge
Description: The impressions of the tooth surface were analysed using scanning electron microscopy (SEM) to investigate changes in the enamel surface topography to determine degree of early stage enamel erosion. Interrogation of the tooth surface via impressions using SEM followed by visual image analysis was used to investigate the enamel surface topography.
  The Images were graded as follows:
  1. - No signs of surface erosive wear (no evidence of the "lock and key" structure)
  2. - Early signs of erosive surface changes
  3. - Mild signs of erosive surface changes (early signs of the "lock and key" structure).
  4. - Moderate signs of erosive surface changes
  5. - Severe signs of erosive surface changes ("lock and key" structure and enamel "pits") X - Not evaluable
Time Frame: Baseline, 30 minutes post dietary acid challenge
Population: The Per Protocol (PP) population was defined as those subjects in the ITT (intent to treat) population who have at least one assessment of efficacy considered unaffected by protocol violation. Assessments of efficacy considered affected by protocol violation were excluded from PP analyses. The primary population was the PP population.
Measure: Median (Full Range); unit: Scores on grading scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
Scores on grading scale | 3.75 (1.917) [0 to 4] | 3.17 (1.882) [0 to 4]
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.2673, Wilcoxon Rank Sum test — P-value was calculated from Wilcoxon Rank Sum test; Median Difference (Final Values) = -0.08, 95% CI 2-sided [-1.0 to 0.0] — Median difference and 95% CI intervals were calculated from the Hodges Lehnmann estimate. Difference was calculated as reference product minus test product

2. Secondary Outcome: Change From Pre-acid Challenge (Baseline) Tooth Impression Grading Score Following 2 Hours Post Acid Challenge.
Description: as for outcome 1
Time Frame: Baseline, 2 hours post acid challenge
Population: The PP population was defined as those subjects in the ITT population who have at least one assessment of efficacy considered unaffected by protocol violation. Assessments of efficacy considered affected by protocol violation were excluded from PP analyses. The primary population was the PP population.
Measure: Median (Full Range); unit: Scores on grading scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
Scores on grading scale | 3.83 [0.0 to 4.0] | 2.33 [0.0 to 3.8]
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.0690, Wilcoxon Rank Sum Test — P-value was calculated from Wilcoxon Rank Sum test; Median Difference (Final Values) = -0.92, 95% CI 2-sided [-1.8 to 0.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Pre-acid Challenge (Baseline) Tooth Impression Grading Score Following 4 Hours Post Acid Challenge
Description: as for outcome 1
Time Frame: Baseline, 4 hours post acid challenge
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on grading scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
Scores on grading scale | 3.17 [0.0 to 4.0] | 1.08 [0.0 to 2.7]
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.0680, Wilcoxon Rank Sum test — P-value was calculated from Wilcoxon Rank Sum test; Median Difference (Final Values) = -1.50, 95% CI 2-sided [-2.7 to 0.0] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Pre-acid Challenge (Baseline) Tooth Impression Grading Score Following 7 Hours Post Acid Challenge
Description: as for outcome 1
Time Frame: Baseline, 7 hours post acid challenge
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on grading scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
Scores on grading scale | 2.58 [0.0 to 4.0] | 0.75 [0.0 to 2.0]
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.0654, Wilcoxon Rank Sum test. — P-value is calculated from Wilcoxon Rank Sum test; Median Difference (Final Values) = -1.83, 95% CI 2-sided [-3.0 to 0.0] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline of Salivary Calcium Concentration at 30 Mins Post Dietary Acid Challenge
Description: Saliva stored at 0 - 20°C was used for determining calcium concentration
Time Frame: Baseline, 30 mins post dietary acid challenge
Population: The PP population was defined as those subjects in the ITT population who have at least one assessment of efficacy considered unaffected by protocol violation. Assessments of efficacy considered affected by protocol violation was excluded from PP analyses. The primary population was the PP population.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
ppm | -12.81 (9.101) | -16.29 (12.041)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.6061, ANCOVA — P value obtained from the ANCOVA analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-6.8 to 4.1] — Difference and 95 % CI obtained from the ANCOVA analysis. Difference was calculated as reference product minus test product

6. Secondary Outcome: Change From Baseline of Salivary Calcium Concentration 7 Hours Post Dietary Acid Challenge
Description: Saliva stored at 0 - 20°C was used for determining calcium concentration
Time Frame: Baseline, 7 hours post dietary acid challenge
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
ppm | 4.38 (10.308) | 0.00 (11.094)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.4080, ANCOVA — P value obtained from the ANCOVA analysis; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-7.9 to 3.3] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline of pH Measurement at 30 Mins Post Dietary Acid Challenge
Description: Saliva stored at 0 - 20°C was used for determining pH
Time Frame: Baseline, 30 mins post dietary acid challenge
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
pH units | -0.71 (0.854) | -0.51 (0.620)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.4611, ANCOVA — P value obtained from the ANCOVA analysis; Median Difference (Final Values) = 0.21, 95% CI 2-sided [-0.4 to 0.8] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Change From Baseline of pH Measurement 7 Hours Post Dietary Acid Challenge
Description: Saliva stored at 0 - 20°C was used for determining pH
Time Frame: Baseline, 7 hours post dietary acid challenge
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
pH units | 0.00 (0.219) | 0.16 (0.569)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.3939, ANCOVA — P value obtained from the ANCOVA analysis; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.1 to 0.3]

9. Secondary Outcome: Change From Baseline in Buffering Capacity at 30 Mins Post Dietary Acid Challenge
Description: Saliva was collected and stored at 0 - 20°C. A Saliva-check Buffer Kit was used to determine the buffer capacity. The colourimetric assay yielded a coloured pattern on a paper diagnostic using a 0-12 scale where 0-5 was deemed to be very low, 6-9 was deemed low and 10-12 was deemed normal-high.
Time Frame: Baseline, 30 mins post dietary acid challenge
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
scores on a scale | -1.81 (3.885) | -1.50 (3.322)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.7829, ANCOVA — P value obtained from the ANCOVA analysis; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-2.2 to 2.8] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Change From Baseline in Buffering Capacity 7 Hours Post Dietary Acid Challenge
Description: as for outcome 9
Time Frame: Baseline, 7 hours post dietary acid challenge
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 16 | 14
scores on a scale | -0.25 (2.463) | -0.36 (2.706)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalent analyses was executed using scale transformation or non-parametric methods; p = 0.9121, ANCOVA — P value obtained from the ANCOVA analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-1.6 to 1.4] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline upto Day 2
Arm/Group | Test Product | Reference Product
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.